CLINICAL TRIAL: NCT01703663
Title: Nasal EPAP for Stroke Patients With Sleep Apnea: a Pilot Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Devin Brown, Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U037625
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Stroke; Obstructive Sleep Apnea
Keywords: Stroke; Sleep Apnea
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea, Obstructive; Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPAP (Experimental): Provent Sleep Apnea Therapy.
  Interventions: Device: EPAP
- control (No Intervention)

INTERVENTIONS:
Device: EPAP
  Other Names: Provent Sleep Apnea Therapy.
  Arms: EPAP

SUMMARY:
Specific aim: To test the effects of nasal expiratory positive airway pressure (EPAP) therapy on sleep apnea severity among patients with recent ischemic stroke.

Hypothesis 1: Ischemic stroke patients with sleep apnea will have less severe sleep apnea, as measured by the apnea-hypopnea index (AHI), with nasal EPAP therapy compared with a control night.

Hypothesis 2: Ischemic stroke patients will have higher mean levels of oxygen saturation with nasal EPAP therapy compared with a control night.

ELIGIBILITY:
Inclusion Criteria:

* adults with an ischemic stroke (including TIA with infarction) within the prior 14 days

Exclusion Criteria:

1. Current use of any transnasal tube (eg dobhoff tube)
2. Current use of CPAP, mechanical ventilation, or supplemental oxygen
3. Known severe breathing disorders including hypercapnic respiratory failure, respiratory muscle weakness, bullous lung disease, bypassed upper airway, pneumothorax, pneumomediastinum
4. Severe heart disease (including severe heart failure)
5. Pathologically low blood pressure
6. An acute upper respiratory (including nasal, sinus or middle ear) inflammation or infection, or perforation of the ear drum
7. Sores, abrasions, or skin or mucosal irritation on or around the nose.
8. Known pregnancy
9. Inability to provide informed consent
10. Use of alpha blockers or short acting nitrates
11. Permanent pacemaker
12. Sustained non-sinus cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin L Brown, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Wheeler NC, Wing JJ, O'Brien LM, Hughes R, Jacobs T, Claflin E, Chervin RD, Brown DL. Expiratory Positive Airway Pressure for Sleep Apnea after Stroke: A Randomized, Crossover Trial. J Clin Sleep Med. 2016 Sep 15;12(9):1233-8. doi: 10.5664/jcsm.6120. PMID 27306393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Some subjects were discharged from the hospital between the first and second night and therefore dropped out.
Groups:
- EPAP Therapy First Night, Then Control Night: During the first night, the subject was assigned to wear EPAP. During the second night, the subject did not wear EPAP (control night). During both nights, sleep disordered breathing was monitored with the WatchPAT device.
- Control Night First Night, EPAP Therapy Second Night: During the first night, the subject was assigned to no EPAP (control night). During the second night, the subject was assigned to wear EPAP. During both nights, sleep disordered breathing was monitored with the WatchPAT device.
Period: First Treatment Period
Arm/Group | EPAP Therapy First Night, Then Control Night | Control Night First Night, EPAP Therapy Second Night
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | EPAP Therapy First Night, Then Control Night | Control Night First Night, EPAP Therapy Second Night
Started | 11 | 8
Completed | 11 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who completed both nights
Arm/Group | All Participants
Number analyzed (Participants) | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [55 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Body mass index, self reported [Median (Inter-Quartile Range); unit: kg/m^2] | 29.1 [26.6 to 33.5]
NIH Stroke Scale [Median (Inter-Quartile Range); unit: units on a scale] — total (range 0-42; 0 is no findings)
  units on a scale | 4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index
Description: Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas and divided by the hours of sleep based on actigraphy. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe. The prespecified primary (absolute) treatment effect is based on the linear repeated measures model.
Time Frame: night 1 and night 2
Measure: Median (Inter-Quartile Range); unit: apneas plus hypopneas per hour
Groups:
- EPAP Night: Raw data from EPAP night (not taking into account period effect).
- Control Night: Raw data from control night (not taking into account period effect).
Arm/Group | EPAP Night | Control Night
Number analyzed (Participants) | 19 | 19
apneas plus hypopneas per hour | 17.1 [13.2 to 26.5] | 25.2 [14.2 to 49.6]
Statistical Analysis 1: Comparison: EPAP Night vs Control Night; Test type: Superiority or Other; p = 0.183, ANOVA; absolute difference = -5.73, 95% CI 2-sided [-14.4 to 2.97]

ADVERSE EVENTS:
Arm/Group | EPAP Night | Control Night
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No